CLINICAL TRIAL: NCT04332952
Title: Damage and Renal Clearance of Glycocalyx in Cardiac Surgery
Acronym: GlycoCarSur
Status: Completed | Type: Observational
Sponsor: Miguel Ayala León (Network)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Sponsor-Investigator, Miguel Ayala León, cardiovascular critical care unit director, Hospital Beneficencia Espanola de Puebla
Organization: Hospital Beneficencia Espanola de Puebla (Network)
Other Study IDs: Cardiologia-002
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Glycocalyx; Cardio-Renal Syndrome
Keywords: Renal clearance; Glycocalyx; Cardiac surgery
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The glycocalyx is a component of the vascular endothelium that currently plays a relevant role in the modified Starling theory.

The manipulation of the heart during cardiac surgery stimulates the release of the natriuretic atrial peptide, which causes endothelial wear in patients undergoing extracorporeal circulation. Dilation of the atrium produces natriuretic atrial peptide, which reduces plasma volume by increasing renal excretion and vascular permeability. The atrial peptide degrades the surface of the coronary endothelium, causing loss of the side cam protein nucleus. This study investigates the relationship between clamping time in cardiac surgery and the clearance of endothelial inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients who underwent cardiac surgery for a single valve change or replacement

Exclusion Criteria:

* Stage 3 renal failure patients
* Patients with a previous diagnosis of hematological malignancy
* Patients undergoing pulmonary valve change surgery.
* Patients undergoing Bentall and Bono surgery.
* Patients Undergoing Coronary Artery Bypass Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the selection criteria undergoing cardiac surgery for a single valve change or replacement.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Extracorporeal circulation time | 2 hours
  Duration of Extracorporeal Circulation in minutes
Aortic clamping time | 2 hours
  Duration of aortic clamping time in minutes
Hyaluronic acid levels in blood before surgery | 30 minutes
  Quantity of hyaluronic acid in blood before surgery
Hyaluronic acid levels in blood after surgery | 30 minutes
  Quantity of hyaluronic acid in blood after surgery
Hyaluronic acid levels in urine before surgery | 30 minutes
  Quantity of hyaluronic acid in urine before surgery
Hyaluronic acid levels in urine after surgery | 30 minutes
  Quantity of hyaluronic acid in urine before surgery
Sydecan -1 levels in blood before surgery | 30 minutes
  Quantity of Sydecan -1 in blood before surgery
Sydecan -1 levels in blood after surgery | 30 minutes
  Quantity of Sydecan -1 in blood after surgery
Sydecan -1 levels in urine before surgery | 30 minutes
  Quantity of Sydecan -1 in urine before surgery
Sydecan -1 levels in urine after surgery | 30 minutes
  Quantity of Sydecan -1 in urine after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beneficencia Española de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No